CLINICAL TRIAL: NCT04746248
Title: The LINO Study - Labor Induction Inpatient and Outpatent: A Pilot- and Feasibility Study of Low-risk Nulliparious Women Using 25 mcg Oral Misoprostol for Labor Induction in an Inpatient and Outpatent Setting in Norway.
Brief Title: Outpatient Labor Induction Using Oral Misoprostol in Norway
Acronym: LINO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Oslo University Hospital (Other); Vestre Viken Hospital Trust (Other)
Responsible Party: Principal Investigator, Mirjam Lukasse, Professor, Oslo Metropolitan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 158844
Record Dates: First submitted 2021-01-25; First posted 2021-02-09 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Induced; Birth; Labor, Induced
Keywords: Labor induction; Induced birth; Outpatient; Oral misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline (No Intervention): The baseline arm includes participants from before the implementation of the outpatient regime. All participants are induced according to the standard inpatient protocol.
- Women choosing to stay at the hospital (Active Comparator): Include women who choose to stay at the hospital after implementing an outpatient alternative.
  Interventions: Other: Inpatient labor induction
- Women choosing to go home (Experimental): Include women who choose the outpatient regime.
  Interventions: Other: Outpatient labor induction

INTERVENTIONS:
Other: Outpatient labor induction — The participants stay at home during til labor induction process and are admitted to hospital at the onset of labor or if a complication occur. Outpatient consultations once a day.
  Arms: Women choosing to go home
Other: Inpatient labor induction — The participants are induced following standard inpatient care
  Arms: Women choosing to stay at the hospital

SUMMARY:
The rate of labor induction has been steadily increasing over the last years, both worldwide and in Norway. Norwegian women are hospitalized when prostaglandins are used to induce labor. In Denmark, a neighboring country to Norway, women have been offered outpatient induction of labor using oral misoprostol for several years.

The overall aim of this study is to investigate if outpatient induction of labor is beneficial in a Norwegian setting. This includes:

1. To investigate the clinical outcomes and feasibility of inducing in an outpatient setting compared to an inpatient setting in Norway
2. To explore low-risk nulliparous women's experiences of labor induction in inpatient and outpatient settings.

This is a non-randomized prospective pilot- and feasibility study, collecting data from electronical records. In addition, the study participants are invited to write a diary during the labor induction process and a questionnaire six weeks postpartum. Eligible patients include low-risk nulliparous women induced with low-dose oral misoprostol.

DETAILED DESCRIPTION:
The labor induction rate in Norway has increased from 10,5 % in 2000 to 26,1 % in 2019. This represents an important shift in the obstetric care, making labor induction one of the most common obstetrical interventions. The increase alters the population being induced, as it now includes more low-risk births compared to 20 years ago. The low risk labor inductions might not require the same repeated cardiotocography and inpatient care before onset of active labor as complicated pregnancies.

In 2017, a 25 μg misoprostol tablet for oral administration was approved for labor induction in the Nordic countries. Oral administration is user friendly, and low-dose orally administrated misoprostol is considered to have a favorable safety profile compared to many other induction methods, with low risk of hyperstimulation.

Despite the widespread knowledge of the importance of women´s labor experience for her future health, this aspect is rarely thoroughly explored in the vast number of studies on labor induction. For outpatient labor induction to work, it must be an alternative women find beneficial, as well as clinicians and the health care system.

Aim

The overall aim of this study is to investigate if outpatient induction of labor is beneficial in a Norwegian setting. This includes:

Study A. To investigate the clinical outcomes and feasibility of inducing in an outpatient setting compared to an inpatient setting in Norway Study B. To explore low-risk nulliparous women's experiences of labor induction in inpatient and outpatient settings.

Design and methods

Study A is a prospective non-randomized multicenter pilot- and feasibility study. Data are collected from the patient's electronical records. Study B is a mixed methods cross-sectional diary study, collecting data from the participants diaries and questionnaire and their electronical records. Both studies include the same participants.

In both the inpatient and outpatient regime, the women are induced with 25 μg misoprostol tablets administrated orally every two hours. Some of the women will be induced using a balloon catheter before misoprostol. In the inpatient regime, cardiotocography (CTG) will be performed according to standard protocol; every 4-6 hours or on indication. In the outpatient protocol, a CTG will be carried out before and after the administration of the first misoprostol. If the CTG is normal and the woman has no contractions, the woman can go home, provided a normal ultrasound scan from the last three weeks. An appointment will be set up no later than 24 hours later for a new CTG and assessment of the induction process and the health of the woman and fetus. If the woman goes home after this consultation, she will return no later than 24 hours later for inpatient labor induction if the labor does not start.

Women choosing the outpatient protocol will receive oral and written information about what they should be aware of and when to contact the maternity ward. They are welcome to contact the maternity ward at any time to seek advice from a midwife with experience in labor induction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy nulliparous women
* A single, healthy fetus in cephalic presentation at gestational age of 37 weeks or more
* Normal pregnancy
* The woman can read and communicate in Norwegian
* No cognitive barriers
* BMI 15,5-39,9
* Reside within one hour from the hospital
* Indication for labor induction is post term pregnancy, uncomplicated pre labor rupture of membranes, maternal wish or other indications determined as low-risk by the attending obstetrician

Exclusion Criteria:

* Known uterine abnormality or previous uterine surgery
* Major maternal medical illness requiring monitoring of mother or fetus in early labor
* Maternal infection
* Pregnancy complications such as preeclampsia, poorly controlled hypertension or medically treated diabetes mellitus
* Active vaginal bleeding characterized as more than bloody show
* Smoking
* Non-reassuring cardiotocography or reduced fetal movement
* Fetal growth EFW < 10th percentile or >90th percentile
* Poly- or oligohydramnios
* Known abnormalities in the placenta or umbilical cord

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The proportion of eligible women selecting outpatient labor induction | up to 18 months
Fetal metabolic acidosis | From delivery and within two hours postpartum
  The proportion of fetal metabolic acidosis
Deliveries outside the hospital | At time of delivery
  The proportion of deliveries outside the hospital in the outpatient versus inpatient induction group

SECONDARY OUTCOMES:
Delivery mode | At the time of delivery
  Mutually exclusive categories, either spontaneous vaginal birth, either instrumental vaginal birth, either operative delivery by cesarean section
Indications for operative delivery | At the time of delivery
  Indications for cesarean delivery or operative vaginal delivery
Uterine rupture | During labor induction or birth
Maternal admission to ICU or maternal death | From start of induction through discharge, normally within 2-4 days after delivery
Maternal hemorrhage (in ml) | During birth and until two hours after delivery
Chorioamnionitis | During birth and until two hours after delivery
  Number of participants with clinical chorioamnionitis
Perineal injury | At the time of delivery
  Perineal third or forth degree lacerations and epiosotomy
Perinatal death | From start of induction until 1 week after delivery
Need for neonatal resuscitation after delivery | Within two hours after delivery
Uterine tachysystole | From start of induction until delivery
Admission to NICU due to birth related issues | From delivery until discharge, usually 2-4 days after delivery, maximum of 1 week postpartum
Apgar score | 1, 5 and 10 minutes after delivery
  Score 0 to 10 where 10 is highest score indicating most vital neonate
Umbilical cord pH and pCO2 | Immediately after delivery
Presence of meconium in amniotic fluid | From start of induction until delivery
Duration of the stages during induction and birth | From start of induction until transfer top postpartum ward
  Time from start of medication to start of active labor, labor duration, duration of hospital stay
Contact with the hospital during the labor induction process | From start of induction until hospital admission
  Counting number of contacts adding up to a total
Misoprostol administration | From start of induction until start of active labor
  Total misoprostol dose, delay of medicament administration
Need for other interventions to induce or augment labor | From start of induction until start of active labor
The experience of labor induction | 6-8 weeks postpartum
  The Experiences of Induction Tool (EXIT), a validated instrument to measure the experiences of labor induction Minimum score per item is 1, maximum is 5, the higher the score the more positive the experience.
The experience of childbirth | 6-8 weeks postpartum
  The Childbirth Experience Questionnaire (CEQ), a validated instrument to measure the experience of childbirth, 4 domains, mean for each domain will be calculated and compared, the higher mean per domain the more positive the birth experience, lowest mean per domain is 1 highest is 4.
Postnatal depression | 6-8 weeks postpartum
  The Edinburgh Postnatal Depression Scale-short version (EPDS-5), Minimum score 0, maximum score 15, cut-off 7 or more The higher the score the more symptoms of depression
The Early Labor Experience | From start of induction until delivery and 6-8 weeks postpartum
  Swedish Early Labor Questionnaire for primiparous women (SWE-ELEQ-PP), a validated instrument to measure measure the experience of early labor, 22 items mean score is calculated, higher score is better experience, minimum score per items is 1 maximum is 5

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Vestre Viken Health Trust, Drammen Hospital, Drammen
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marsdal KE, Sorbye IK, Bernitz S, Adan N, Grodal EB, Jacobsen AF, Lukasse M. Clinical outcomes and feasibility of implementing outpatient labor induction with misoprostol: A prospective cohort study. Acta Obstet Gynecol Scand. 2025 Apr;104(4):647-657. doi: 10.1111/aogs.15029. Epub 2025 Jan 29. PMID 39878306